CLINICAL TRIAL: NCT06314048
Title: Teamwork, Targets, Technology, and Tight Control in Newly Diagnosed Pediatric T1D: 4T Sustainability Program.
Brief Title: 4T Sustainability Program
Status: Enrolling by invitation | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, David Maahs, Chief of Pediatric Endocrinology, Stanford University
Other Study IDs: 74212
Record Dates: First submitted 2024-02-15; First posted 2024-03-15 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Type1diabetes
Keywords: Pediatric; Type 1 Diabetes; Continuous Glucose Monitor; Remote Patient Monitoring; Patient Reported Outcomes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Standard of Care - CGM and RPM: 1. Implement the 4T program as standard of care at Stanford Diabetes clinics, including Continuous Glucose Monitoring (CGM) and Remote Patient Monitoring (RPM) within the first 30 days after T1D diagnosis to reduce the rise in HbA1c trajectory observed 4-12 months post-diagnosis.
  Interventions: Other: CGM and RPM

INTERVENTIONS:
Other: CGM and RPM — 1. Implement the 4T program as standard of care at Stanford Diabetes clinics, including Continuous Glucose Monitoring (CGM) and Remote Patient Monitoring (RPM) within the first 30 days after T1D diagnosis to reduce the rise in HbA1c trajectory observed 4-12 months post-diagnosis.

SUMMARY:
The goal of the 4T program is to implement proven methods and emerging diabetes technology into clinical practice to sustain tight glucose control from the onset of type 1 diabetes (T1D) and optimize patient-reported and psychosocial outcomes. The investigators will expand the 4T (Teamwork, Targets, Technology, and Tight Control) program to all patients seen at Stanford Pediatric Diabetes Endocrinology as the standard of care. Disseminating the 4T program as the standard of care will optimize the benefits of diabetes technology by lowering HbA1c, improving PROs, and reducing disparities.

DETAILED DESCRIPTION:
The investigators propose a multi-disciplinary diabetes team approach to utilize existing and emerging diabetes technologies and education strategies to implement scalable diabetes care with the goal of maintaining tight control for newly diagnosed Pediatric T1D patients. Successful T1D care is more than glucose control; the 4T program will closely monitor psychosocial and patient-reported outcomes (PROs) through the established psychosocial screening and treatment program. The 4T program will utilize automated approaches to analyze glucose profiles developed in conjunction with the Stanford SURF (Systems Utilization Research For Stanford Medicine) team. The 4T program will tailor intervention to those patients most in need of team support employing a broad range of behavioral and technology supports, strengths of the Stanford Pediatric Diabetes program. The 4T program approach more precisely adapts care to patient needs and optimizes glucose and psychosocial outcomes.

Therefore, the investigators propose to expand the diabetes team approach (Teamwork, Targets, and Technology for Tight Control: 4T), which utilizes existing diabetes technologies and education strategies to implement and standardize goal-oriented diabetes care for newly diagnosed pediatric T1D patients, to a standard of care program at Stanford pediatric diabetes clinics. The Stanford diabetes team has revised the diabetes education approach to set clear and tighter targets at new-onset through the early phase of T1D and to be aggressive with the intensification of control as insulin needs and care demands increase. The 4T Sustainability program will further standardize T1D team care while allowing for personalization based on patient/family needs with the goal of optimizing glucose and psychosocial outcomes. (NOTE: the current protocol [IRB #52812] focuses on early initiation of CGM as the key technology for glucose monitoring. The 4T program is designed to be flexible to incorporate emerging technologies as they become available for patient care. For example, automated insulin delivery systems will be supported as part of the program). To make the 4T Sustainability Program a true standard of care program, remote patient monitoring (RPM) of the CGM data and CDCES-tailored patient contacts will be billed using RPM billing codes. These RPM billing codes have received hospital compliance approval, and billing workflows will be available in LPCH EPIC.

Personalized Goals and Automated Identification for Need for Insulin Changes in New Onsets: Data collected by continuous glucose monitoring (CGM) can improve the quality of patient care; facilitate the use of telemedicine to reduce costs and improve convenience; and improve the understanding of how daily behaviors shape long-term outcomes.

Modern Electronic Health Records (EHRs) can potentially be used to reduce the workload necessary to care for patients; reduce error rates by automating alerts; and facilitate continuous evaluation and improvement of provider adherence to best-practices. To be practical and scalable, these systems must provide actionable information and require relatively few inputs. The investigators have developed stand-alone tools that analyze CGM time series data to set personalized care goals and to determine when glucose values increase, or insulin dose adjustments and other care adaptations are required. To allow Stanford and the broader community to realize the full potential of such tools, the investigators will implement and refine their use in our clinics:

1. Implement and refine analytical methods and software tools to interpret and improve the quality of time-series CGM data, set personalized goals, and generate automated notifications for care providers.
2. A data-driven intervention to improve long-term outcomes for early onset patients including a hospital- server-based monitoring system to evaluate the intervention. [Note: identification is the goal of the system and medical advice will be solely given by trained healthcare professionals.]

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria includes all youth with new onset T1D seen in the Stanford/Lucile Packard Children's Hospital ages 6 months-21 years of age. The program will also be offered to pediatric patients with existing T1D who wear a CGM or want to start a CGM and receive RPM. We intend to include all possible patients with the goal of maximizing generalizability of the results and 4T program. (NOTE: We will include children and families who speak all languages using the Stanford interpreter services so as to have the greatest generalizability of the research. Questionnaires will only be given to English and Spanish speakers.)

* All individuals with a T1D diagnosis seen at the Stanford Children's Diabetes Clinic
* Individuals who plan to receive follow-up care at the Stanford Children's Diabetes Clinic
* Individuals who agree to wear a CGM that will connect to the RPM-care model
* Age: six months to < 21 years of age
* Patient or guardian must own and operate a compatible smart device/phone to send data from the CGM into the HIPAA-compliant RPM-care model for data analysis and review by a care team member.

  * Dr. Maahs and Pediatric Endocrinology have philanthropic funds available to purchase compatible smart devices for participants who do not have a compatible smart device/phone.

Exclusion Criteria:

* Diabetes diagnosis other than T1D
* Individuals with the intention of obtaining diabetes care at another clinic
* Individuals who do not consent to CGM use, CGM data integration, remote monitoring
* Individuals > 21 years of age

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients seen at Stanford Children's Diabetes Clinic diagnosed with Type 1 Diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c trajectory observed 4-12 months post-diagnosis | 4-12 months post TID diagnosis
  Implement 4T program as standard of care, including Continuous Glucose Monitoring (CGM) and Remote Patient Monitoring (RPM) within the first 30 days after T1D diagnosis to reduce the rise in HbA1c trajectory observed 4-12 months post-diagnosis.To address Aim 1, the investigators will use generalized linear mixed effects regression techniques that allows for two piecewise linear slopes of HbA1c levels to be estimated from diagnosis to 4 months and from 4 to 12 months post-diagnosis to determine the effect of the 4T diabetes intervention on changes in HbA1c between 4- and 12-months post-diagnosis and compare observed increases to those in our internal and external contemporaneous controls via separate models. Each mixed effects model will include a subject-specific random effect to account for the correlation of HbA1c within a person over time, and these models will be adjusted for sex, age, ethnicity, and insurance type at diagnosis.
Diabetes distress measured at baseline and 12 months post-diagnosis. | baseline and 12 months post Type 1 Diabetes diagnosis
  The investigators will utilize generalized linear mixed effects models to address Aim 2. More specifically, the investigators will regress diabetes distress index on use of CGM. Such a model will include a subject-specific random effect and an indicator of whether the patient utilized CGM technologies.
  Assuming the ratio of using CGM technology is 0.6 and SD of diabetes distress score is 3, we have 90% power to detect a two-unit reduction on mean diabetes distress score.

CONTACTS AND LOCATIONS:
Overall Officials: David M Maahs, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No